CLINICAL TRIAL: NCT01654159
Title: Evaluating Subjective and Objective Performance of Instrumentation Used and Devices Implanted in Cataract Surgery
Brief Title: Assessment of Visual Function and Optics in Intraocular Lenses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOL2012
Record Dates: First submitted 2012-07-17; First posted 2012-07-31 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cataract
Keywords: intraocular lenses; evaluation; cataract
MeSH Terms: conditions — Cataract | interventions — Multifocal Intraocular Lenses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Monofocal (Placebo Comparator): Monofocal IOL Implant
  Manufacturers of IOLs used as monofocal comparator are Alcon, AMO, Bausch and Lomb, Lenstec, Oculentis, Ophthec, Physiol and Zeiss
  Interventions: Procedure: Monofocal IOL
- Multifocal (Experimental): Multifocal IOL
  Manufacturers of multifocal IOLs under investigation are Alcon, AMO, Bausch and Lomb, Lenstec, Oculentis, Ophthec, Physiol and Zeiss
  Interventions: Procedure: Multifocal IOL
- Toric (Experimental): Toric IOL
  Manufacturers of toric IOLs under investigation are Alcon, AMO, Bausch and Lomb, Lenstec, Oculentis, Ophthec, Physiol and Zeiss
  Interventions: Procedure: Toric IOL

INTERVENTIONS:
Procedure: Monofocal IOL — Monofocal Intraocular lens will be implanted
  Other Names: Alcon AMO B&L Lenstec Oculentis Ophthec Physiol & Zeiss
  Arms: Monofocal
Procedure: Multifocal IOL — Multifocal IOL will be implanted
  Arms: Multifocal
Procedure: Toric IOL — Toric IOLS will be implanted
  Arms: Toric

SUMMARY:
The main objective of this research is to assess visual function and optical performance of CE marked, implanted intraocular lenses to understand the individual factors that affect their performance and how these may be improved in future designs and to evaluate measurement techniques.

All outcome measures will be captured 3-6 months after surgery

DETAILED DESCRIPTION:
A cataract occurs when the natural lens of the eye, which plays a major role in the focusing of light and production of sharp visual images, becomes cloudy and hardens, resulting in a loss of visual function. Left untreated, cataracts can cause preventable blindness. During cataract surgery the natural lens is removed and a man-made intraocular lens (IOL) is implanted in its place.

IOL technology has advanced significantly in recent years and as a result the main goal of cataract surgery is no longer simply the successful removal of the cloudy lens and restoration of vision. Providing patients with the best possible refractive outcome and the best possible visual quality is now much more important when assessing surgery outcomes.

Aspheric, multifocal and accommodating IOLs are among the new designs developed to improve visual outcome after cataract surgery. In order to assess the effectiveness of these designs, visual function needs to be evaluated both objectively and subjectively following their implantation. Such evaluation allows the continued evolution of these IOL designs towards optimum. This proposed research study, which aims to assess the visual function and optical performance of new CE marked IOLs after implantation, could significantly contribute to the enhancement and development of improved IOL designs in the future.

We have successfully conducted similar patient trials for the past 5 years. As new IOL designs are constantly being developed, approved and CE marked, this type of research study will always have the potential to offer new information that is not currently available and has not previously been assessed or published and could contribute towards improved IOL designs in the future.

All outcome measures will be captured 3-6 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Subjects age between 40-85 years, may be either male or female, and may be of any race (as cataracts rarely occur before the age of 40 and above 85 other ocular pathology is common).
* Subjects requiring cataract surgery.
* Potential for best corrected visual acuity of 6/12 or better (as visual function in these patients will be affected by ocular pathology).
* Subjects with clear intraocular media other than cataract (as assessing cataract).
* General physical and mental condition allowing participation in current study.
* Subjects willing to participate as evidenced by signing the written informed

Exclusion Criteria:

* Prior surgery on the selected eye
* Previous uveitis or trauma to the selected eye, anterior or posterior synechiae
* Potential for best corrected visual acuity worse than 6/12 (since this may indicate other causes of ocular pathology)
* Partial or total paralysis, Parkinsons syndrome, cerebrovascular accident or other condition that could impact on the results of the study
* Subject over 85 years of age (ocular pathology more common in this age group)
* Subjects without adequate physical and mental capacity to enable participation in the study
* Subject unwilling to participate
* Systemic or topical medication known to influence visual function measures

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Unaided distance and near vision | Measured at 3-6 months after surgery
  Visual Acuity (logMAR)

SECONDARY OUTCOMES:
Patient Satisfaction | Measured at 3-6 months after surgery
  NAVQ score
Residual refraction | Measured at 3-6 months after surgery
  Autorefraction / subjective refraction
Aberrations | Measured at 3-6 months after surgery
  Aberrometry
Corrected distance and near acuity | Measured at 3-6 months after surgery
  Acuity (logMAR)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Shah, FRCS, Principal Investigator — Birmingham Midland Eye Centre
Locations (1):
- Birmingham Midland Eye Centre, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data collaboration will be considered on request